CLINICAL TRIAL: NCT04186715
Title: The Effect of Vestibular Transoral Endoscopic Thyroidectomy on Cerebral Regional Oxygen Saturation: Comparison With Open Thyroidectomy
Brief Title: Near Infrared Spectroscopy in Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaEAH01
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2019-11

CONDITIONS: Thyroidectomy; Near-infrared Spectroscopy
Keywords: TOETVA; Thyroidectomy; near-infrared spectroscopy
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TOETVA: The demographic data of the patients undergoing TOETVA surgery will be recorded. Then, blood pressure, pulse pressure, pulse oximeter, end-tidal carbon dioxide, right and left cerebral regional oxygen values in the operation room will be recorded at certain intervals. It will also be recorded if complications develop.
  Interventions: Device: Near-infrared spectroscopy
- Open thyroidectomy: The demographic data of the patients undergoing open thyroidectomy surgery will be recorded. Then, blood pressure, pulse pressure, pulse oximeter, end-tidal carbon dioxide, right and left cerebral regional oxygen values in the operation room will be recorded at certain intervals. It will also be recorded if complications develop.
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — The Near-infrared spectroscopy probes will be placed in the frontal region.

SUMMARY:
Thyroidectomy operations have traditionally been performed as open surgery. However, the scarring that occurs in the patient leads to cosmetic problems, especially in young women. Today, as a result of the development of minimally invasive surgical techniques, the number of natural orifice transluminal endoscopic surgeries (NOTES) is increasing. Surgical scars are avoided by using natural pathways such as the mouth, urethra, vagina or anus. Transoral endoscopic thyroidectomy (TOETVA) with vestibular approach, a form of NOTES, was first performed in 2011. In this method, the operation is performed through three ports entered near the gingiva-buccal sulcus. TOETVA surgeries are performed with an insufflation pressure of 6 mmHg in the neck region. No studies are examining the effects of this pressure on the blood vessels in the neck region on the blood supply to the brain tissue. Therefore, the investigators aim to compare cases operated using open thyroidectomy or TOETVA method by measuring cerebral regional tissue saturation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

Exclusion Criteria:

* Patients with neck surgery.
* Patients who received radiotherapy to the neck region.
* Patients with cerebrovascular or neurological disease.
* Patients who underwent open surgery during the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to our Institute for thyroidectomy.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
cerebral regional oxygen saturation in TOETVA and open thyroidectomy | Before induction
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in TOETVA and open thyroidectomy | 10 minutes after induction
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in TOETVA and open thyroidectomy | 5 minutes after operation position
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in TOETVA | 10 minutes after insufflation
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in TOETVA | 10 minutes after desufflation
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in open thyroidectomy | 10 minutes after platysma incision
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in open thyroidectomy | 10 minutes after the closing of the platysma
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.
cerebral regional oxygen saturation in TOETVA and open thyroidectomy | Through operation completion, an average of 4 hours
  The values obtained from the right and left frontal region will be recorded through the near Infrared Spectroscopy probes.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan OZYURT, MD, Principal Investigator — University of Health Sciences, Antalya Training and Research Hospital
Locations (1):
- University of Health Sciences, Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No